CLINICAL TRIAL: NCT03280836
Title: Women In Steady Exercise Research - Neoadjuvant Exercise Trial
Brief Title: Exercise Program in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Acronym: WISER-NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5517
Record Dates: First submitted 2017-08-31; First posted 2017-09-13 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasm; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are randomized to the intervention or control arm.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): We ask that participants in the control arm do not start an exercise program.
- Exercise (Experimental): Participants in the experimental arm will be asked to complete the exercise intervention with 80% or greater adherence.
  Participants will work towards the goal of 75 or more minutes a week of moderate to vigorous exercise. Participants are provided an exercise toolkit and directed on exercise progression based on personal fitness level.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — All participants randomized to the intervention group will be asked to keep an exercise log with the date, time, average heart rate obtained from a heart rate monitor, duration of workout and stretching, and any comments regarding the workout. Participants will be instructed to bring workout logs to infusion sessions for review. Participants will also wear a Polar Heart Rate monitor (US model RS400, Polar Electro Inc., Lake Success, NY) during exercise to monitor exercise intensity.
  The aerobic exercise intervention will work toward the target of 75 minutes physical activity per week at 60%-85% of baseline VO2max.
  Arms: Exercise

SUMMARY:
The investigators seek to conduct a home based exercise intervention in breast cancer patients whom elect to undergo neoadjuvant chemotherapy. The primary aim of the study is to determine whether breast cancer patients can be enrolled, randomized, retained, and comply with exercise program; and, the feasibility of acquiring, managing and analyzing clinical data.

DETAILED DESCRIPTION:
Several national and international agencies recommend exercise participation for all persons following a cancer diagnosis. The current evidence suggests that aerobic exercise training is safe during primary adjuvant therapy and improves cardiopulmonary function and patient related outcomes. Cardiopulmonary fitness is highly predictive of overall and cardiovascular specific mortality in women. Specifically, an increase in cardiopulmonary fitness of approximately 10% has been associated with a 19% reduction in risk for CV mortality. This is important as breast cancer patients already present at diagnosis with 31% lower cardiopulmonary fitness levels compared to healthy age-matched women. This enhanced risk for cardiovascular mortality in breast cancer patients is further compounded by cardiotoxic chemotherapy, which causes permanent cardiac damage. Few studies have tested the efficacy of exercise prescriptions that incorporate high intensity aerobic exercise training in cancer patients, especially those receiving chemotherapy. Therefore, the investigators seek to conduct an at home aerobic exercise training intervention in breast cancer patients whom elect to undergo neoadjuvant chemotherapy

ELIGIBILITY:
3.1 Inclusion Criteria

* Women with a breast cancer diagnosis (Stage I-IIIC)
* Sedentary (< 75 min/wk of moderate intensity exercise over the past month)
* No previous history of anthracycline based chemotherapy
* Absence of heart disease (clinical diagnosis of coronary artery disease, arrhythmias, congenital heart defects, dilated cardiomyopathy, or valvular heart disease)
* Absence of contraindications for neoadjuvant chemotherapy
* Scheduled to receive neoadjuvant chemotherapy
* Primary attending oncologist approval

3.2 Exclusion Criteria

* Absolute contraindications for exercise stress testing

  * acute myocardial infarction (3-5 days)
  * unstable angina
  * uncontrolled arrhythmias causing symptoms or hemodynamic compromise
  * syncope
  * acute endocarditis
  * acute myocarditis or pericarditis
  * uncontrolled heart failure
  * acute pulmonary embolus or pulmonary infarction
  * thrombosis of lower extremities
  * suspected dissecting aneurysm
  * uncontrolled asthma
  * pulmonary edema
  * room air desaturation at rest ≤85%
  * respiratory failure
  * acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
  * mental impairment leading to inability to cooperate
  * decisional impairment
* Non-English speaking
* Women only diagnosed with ductal carcinoma in situ
* Women diagnosed with stage 4 metastatic breast cancer
* Pregnant women
* Men
* Children

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Sturgeon, PhD, Principal Investigator — Assistant Professor, Penn State
Locations (2):
- United States (2):
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sturgeon KM, Smith AM, Federici EH, Kodali N, Kessler R, Wyluda E, Cream LV, Ky B, Schmitz KH. Feasibility of a tailored home-based exercise intervention during neoadjuvant chemotherapy in breast cancer patients. BMC Sports Sci Med Rehabil. 2022 Feb 25;14(1):31. doi: 10.1186/s13102-022-00420-6. PMID 35216638

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: Participants in the experimental arm will be asked to complete the exercise intervention with 80% or greater adherence.
  Participants will work towards the goal of 75 or more minutes a week of moderate to vigorous exercise. Participants are provided an exercise toolkit and directed on exercise progression based on personal fitness level.
  Exercise: All participants randomized to the intervention group will be asked to keep an exercise log with the date, time, average heart rate obtained from a heart rate monitor, duration of workout and stretching, and any comments regarding the workout. Participants will be instructed to bring workout logs to infusion sessions for review. Participants will also wear a Polar Heart Rate monitor (US model RS400, Polar Electro Inc., Lake Success, NY) during exercise to monitor exercise intensity.
  The aerobic exercise intervention will work toward the target of 75 minutes physical activity per week at 60%-85% of baseline VO2max.
Period: Overall Study
Arm/Group | Control | Exercise
Started | 10 | 9
Completed | 9 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Exercise | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (9.5) | 47.0 (11.7) | 49.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: Percent of Eligible Patients That Provide Consent and Are Enrolled in the Study.
Description: Acceptability of the study will be assessed by documenting the percent of eligible patients that provide consent and are enrolled in the study.
Time Frame: 4 weeks
Population: * Female breast cancer patients (Stage I-IIIC)
  * Sedentary
  * No previous history of anthracycline based chemotherapy
  * Absence of heart disease
  * Absence of contraindications for neoadjuvant chemotherapy
  * Scheduled to receive neoadjuvant chemotherapy
  * Primary attending oncologist approval
  * English speaking
  * Absence of contraindications for exercise stress testing
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Individuals: The target population that is eligible for the study is:
  * Women with a breast cancer diagnosis (Stage I-IIIC)
  * Sedentary (< 75 min/wk of moderate intensity exercise over the past month)
  * No previous history of anthracycline based chemotherapy
  * Absence of heart disease (clinical diagnosis of coronary artery disease, arrhythmias, congenital heart defects, dilated cardiomyopathy, or valvular heart disease)
  * Absence of contraindications for neoadjuvant chemotherapy
  * Scheduled to receive neoadjuvant chemotherapy
  * Primary attending oncologist approval
  * English speaking
  * Absence of contraindications to exercise stress testing
Arm/Group | All Eligible Individuals
Number analyzed (Participants) | 74
Participants | 19

2. Primary Outcome: Participant Adherence to the Exercise Intervention
Description: Tolerability was defined for each intervention exercise training phase by the percent of weekly exercise minutes completed at the prescribed exercise intensity according to the patient's heart rate monitor.
Time Frame: Introduction phase of prescribed exercise training (weeks 1-4), intermediate phase of prescribed exercise training (weeks 5-11), maintenance phase of prescribed exercise training (weeks 12-chemotherapy completion)
Population: The control group was not given heart rate monitors or an exercise prescription.
Measure: Mean (Standard Error); unit: % exercise time at prescribed heart rate
Arm/Group | Control | Exercise
Number analyzed (Participants) | 0 | 6
% exercise time at prescribed heart rate
  Introduction phase |  | 72.7 (11.5)
  Intermediate phase |  | 61.0 (5.0)
  Maintenance phase |  | 23.7 (7.1)

3. Primary Outcome: Change in Cardiopulmonary Fitness Level From Baseline to the Window Following Chemotherapy Completion and Before Surgical Resection
Description: Expired gas analysis (oxygen used by the body) during a submaximal treadmill exercise test determined cardiopulmonary fitness. Change between baseline and the window following chemotherapy completion and before surgical resection, was calculated as the value at the test conducted in the window following chemotherapy completion and before surgical resection minus the value at the test conducted at baseline.
Time Frame: Baseline and the window following chemotherapy completion and before surgical resection (no longer than 26 weeks from baseline)
Population: Patients that withdrew, were lost to follow up, or developed treatment-induced contraindications to exercise testing, are not included in the analysis population.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Control | Exercise
Number analyzed (Participants) | 6 | 7
ml/kg/min | -27.5 (7.4) | -1.0 (13.2)

ADVERSE EVENTS:
Time Frame: Approximately 9 months, from consent to final testing.
Description: Systematic review of EMR for serious adverse events, systematic use of injury history questionnaire at follow up testing. The injury history questionnaire contains self-report for all adverse events that are specific and non-specific to exercise training. The "at Risk" population for "Other (Not Including Serious) Adverse Events" is reflective of women that completed the questionnaire at follow up.
Arm/Group | Control | Exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/10 | 5/9
Other Adverse Events (participants affected / at risk) | 4/7 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | Exercise (N=9)
Thrombosis/embolism (Vascular disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=7) | Exercise (N=7)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was closed to recruitment at n=19, 1 patient short of anticipated enrollment (n=20) due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03280836/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT03280836/ICF_001.pdf